CLINICAL TRIAL: NCT07216170
Title: REVascularization In Large VEssel Occlusion for Acute Ischemic Stroke
Acronym: REVIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TER-CL-5000
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Intracranial large vessel occlusive disease; Revascularization; Large bore catheter; Mechanical thrombectomy; Aspiration; SOFIA®; Direct Aspiration
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SOFIA Flow 88 Aspiration Catheter (Experimental)
  Interventions: Device: SOFIA Flow 88 Aspiration Catheter

INTERVENTIONS:
Device: SOFIA Flow 88 Aspiration Catheter — The investigational device is the SOFIA Flow 88 Aspiration Catheter with the MV Flow Aspiration Pump and MicroVention Tubing Kit and is intended for use in the revascularization of patients with acute ischemic stroke secondary to intracranial large vessel occlusive disease (within the internal carotid, middle cerebral - M1 segment) within 8 hours of symptom onset.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the SOFIA Flow 88 Aspiration Catheter for treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
The investigation is a prospective, single-arm, multi-center clinical study. The study will be conducted in up to 40 investigational sites in the US, Canada, and Europe. This study will enroll up to 200 subjects, with a maximum enrollment of 30 subjects per site.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years on the date of consent
2. National Institutes of Health Stroke Score (NIHSS) ≥6
3. Alberta Stroke Program Early CT Score (ASPECTS) ≥6 assessed within 120 minutes before arterial access, defined by either baseline non-contrast computed tomography (NCCT) or baseline diffusion-weighted magnetic resonance imaging (DW-MRI)
4. Angiographically suitable for endovascular intervention and the interventionalist estimates that arterial access can be achieved within 8 hours from time last known well
5. Independent status immediately pre-stroke defined as ability to perform all activities of daily living as defined by mRS 0-1
6. Large vessel occlusion of the intracranial internal carotid artery (ICA), middle cerebral artery (MCA) M1 segment technically accessible, as assessed during the index procedure, using a SOFIA Flow 88 Aspiration Catheter
7. Subject or legally authorized representative (LAR) is willing and able to provide informed consent, as evidenced by signing and dating the IRB-approved informed consent form prior to initiation of any study-specific procedures
8. Willing and able to comply with the protocol-specified procedures and assessments

Exclusion Criteria:

1. Any intracranial hemorrhage at baseline
2. Previous stroke within 90 days
3. Female who is pregnant or lactating or has a positive pregnancy test at time of admission
4. Arterial occlusive lesion is not technically amenable to recanalization, as assessed during the index procedure, using a SOFIA Flow 88 Aspiration Catheter (e.g., an extracranial carotid lesion prevents access, evidence of carotid dissection)
5. Clinical symptoms or non-invasive imaging suggestive of or confirming bilateral stroke or stroke in multiple territories defined as multiple large vessel occlusions (e.g., bilateral proximal MCA occlusions)
6. Comorbid illness that would confound the neurological or functional evaluation or is severe enough (e.g., metastatic cancer, severe congestive heart failure) such that life expectancy is <1 year or the 90-day outcome is likely to be determined by the comorbid illness
7. Any contraindication to endovascular thrombectomy, such as a known history of severe contrast allergy or absolute contraindication to iodinated contrast
8. Participation in another clinical trial involving an investigational mechanical device (subjects may be co-enrolled in a registry study where there is no investigational treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of all symptomatic intracranial hemorrhage (sICH) | 24 hours post-procedure
Reperfusion success | During procedure
  Defined as independent core laboratory adjudicated modified thrombolysis in cerebral infarction (mTICI)/expanded thrombolysis in cerebral infarction (eTICI) ≥2b flow, using the SOFIA Flow 88 Aspiration Catheter only within ≤ 3 passes and without additional intraprocedural mechanical thrombectomy devices or intra-arterial thrombolytic therapy.

SECONDARY OUTCOMES:
Reperfusion success (defined as independent core laboratory adjudicated mTICI/eTICI ≥2b flow) | During procedure
Time from arterial access to achieve mTICI/eTICI ≥2b | During procedure
Incidence of mTICI/eTICI 3 reperfusion | During procedure
Incidence of mTICI/eTICI ≥2c reperfusion | During procedure
Incidence of mTICI/eTICI ≥2b reperfusion achieved with first pass of the SOFIA Flow 88 Aspiration Catheter | During procedure
Incidence of mTICI/eTICI ≥2c reperfusion achieved with first pass of the SOFIA Flow 88 Aspiration Catheter | During procedure
Incidence of functional independence (modified Rankin scale (mRS) ≤2) | 90-days follow-up
Mortality | 90 days post-procedure
Incidence of intracranial hemorrhage (ICH) | 24 hours post-procedure
Incidence of Embolization to New Territory | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hill, MD, MSc, Principal Investigator — University of Calgary & Foothills Medical Centre; Charles Matouk, MD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No